CLINICAL TRIAL: NCT06390384
Title: Prevention Programme for Improvement of Well-being and Level of Participation in Adolescents With Enhanced Psychiatric Burden in the School Environment.
Acronym: STEPS@SCHOOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STEPS@SCHOOL
Record Dates: First submitted 2024-04-11; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Blended-care Counselling; Digital and Mental Literacy Training; App STEPS
Keywords: eMental health; digital health; blended care treatment; students at risk in schools; psychiatric disorders; adolescents
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The intervention is a implementation of a weekly psychological counseling for psychiatric problems via videoconference combined with an additionally digital support using a well-established mobile treatment system STEPS®. The intervention will include: 1) digital and mental literacy training for children, parents and teachers in the school; 2) weekly counselling over 6 weeks via videoconference for adolescents and their parents; 3) blinded-care use of the mobile treatment system STEPS®.
  Control condition (Treatment as Usual) includes the implementation of the digital and mental literacy training, however, no weekly counselling by the team of the clinic and no blinded-care use of the mobile treatment system STEPS®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): blinded-care counselling + App STEPS + digital and mental literacy training
  Interventions: Other: blinded-care counselling; Other: App STEPS; Other: digital and mental literacy training
- TAU group (Treatment as Usual) (No Intervention): digital and mental literacy training

INTERVENTIONS:
Other: blinded-care counselling — The intervention is a implementation of a weekly psychological counseling for psychiatric problems via videoconference combined with an additionally digital support using a well-established mobile treatment system STEPS®. The intervention will include: 2) weekly counselling over 6 weeks via videoconference for adolescents and their parents.
  The counselling will be provided by experienced psychologists as employers of the Clinic of Child and Adolescent Psychiatry, RWTH Aachen University, the counselling will be supervised by the leading psychologist of the clinic. The counselling will include psychoeducative elements about psychological and psychosocial problems, behavioral interventions from cognitive-behavioral therapy, psychological techniques for better coping with stress, different therapeutic tasks such as fear exposure, activation exercises e.c. The students will be instructed to use the mobile treatment system STEPS in order to continue therapy at home.
  Arms: Intervention group
Other: App STEPS — The intervention is a implementation of a weekly psychological counseling for psychiatric problems via videoconference combined with an additionally digital support using a well-established mobile treatment system STEPS®. The intervention will include: 3) blinded-care use of the mobile treatment system STEPS®.
  This is transdiagnostic digital treatment system which consists of a students front-end as an App and a therapist front-end as an online platform. The App and the platform are connected to each other. In such a way, an effective data transter (for example, symptom evaluation by the student and tasks and requests by the therapist), direct communication between a student and a therapist, as well as registration of emergency situation, are possible.
  Arms: Intervention group
Other: digital and mental literacy training — The intervention is a implementation of a weekly psychological counseling for psychiatric problems via videoconference combined with an additionally digital support using a well-established mobile treatment system STEPS®.
  The intervention will include: 1) digital and mental literacy training for children, parents and teachers in the school.
  This training program (4 weeks, 8 session a 2 lesson units, 2 sessions a week) includes information about rules and functions by using mobile applications, safety aspects of personal data, risks associated with data sharing, sexing and cybergrooming, managing social media, handling with fake news, influence of social media on mental health, forms of digital violence and strategies to cope with them.
  Arms: Intervention group

SUMMARY:
The objectives of this two-arm phase-IIa randomized, controlled study are:

* to prove whether the combination of a clinic-guided personal counseling with a therapy-assistive digital support (blinded care approach) and a training of digital and mental health literacy is superior to a teacher-guided training of digital and mental health literacy only (treatment as usual) concerning the reduction of psychiatric burden in adolescents.
* to improve the well-being and level of participation in adolescents at risk for psychiatric disorders.
* to reduce the expression of psychiatric symptoms in adolescents with enhanced psychiatric burden.
* to test whether the combination of a clinic-guided personal counseling with a therapy-assistive digital support is well accepted by students, their parents, and teachers.
* to identify individual factors predicting the improvement of well-being and level of participation in adolescents as well as the acceptance of the prevention program in all subjects involved (students, parents, teachers, psychologists).
* to investigate whether the clinic-guided personal counseling with a therapy-assistive digital support causes reduction of primary and secondary costs in the psychosocial support system and represents an economic advantage.

DETAILED DESCRIPTION:
The objectives of this two-arm phase-IIa randomized, controlled study are:

* to prove whether the combination of a clinic-guided personal counseling with a therapy-assistive digital support (blinded care approach) and a training of digital and mental health literacy is superior to a teacher-guided training of digital and mental health literacy only (treatment as usual) concerning the reduction of psychiatric burden in adolescents.
* to improve the well-being and level of participation in adolescents at risk for psychiatric disorders.
* to reduce the expression of psychiatric symptoms in adolescents with enhanced psychiatric burden.
* to test whether the combination of a clinic-guided personal counseling with a therapy-assistive digital support is well accepted by students, their parents, and teachers.
* to identify individual factors predicting the improvement of well-being and level of participation in adolescents as well as the acceptance of the prevention program in all subjects involved (students, parents, teachers, psychologists).
* to investigate whether the clinic-guided personal counseling with a therapy-assistive digital support causes reduction of primary and secondary costs in the psychosocial support system and represents an economic advantage.

The STEPS@SCHOOL clinical study is a two-arm parallel group phase-IIa randomized, non-blinded, controlled study with four measurement points (T1: confirming the risk status/checking inclusion criteria/informed consent; T2: baseline assessment and randomization prior to start of intervention; T3: post intervention assessment; T4: three months follow-up). The study will prove whether the combination of a clinic-guided personal counseling with a therapy-assistive digital support (first arm) is superior to a teacher-guided digital preventive platform with stand-alone digital applications (second arm, described as treatment as usual) concerning the reduction of psychiatric burden in adolescents. To prove this objective, a comparison between two groups (treatment of approval vs. treatment as usual) is necessary.

The intervention is a implementation of a weekly psychological counseling for psychiatric problems via videoconference combined with an additionally digital support using a well-established mobile treatment system STEPS®. The intervention will include: 1) digital and mental literacy training for children, parents and teachers in the school; 2) weekly counselling over 6 weeks via videoconference for adolescents and their parents; 3) blinded-care use of the mobile treatment system STEPS®.

Control condition (Treatment as Usual) includes the implementation of the digital and mental literacy training, however, no weekly counselling by the team of the clinic and no blinded-care use of the mobile treatment system STEPS®.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents of both genders (w : m = 1 : 1) aged from 10 to 14 years
* Psychiatric symptoms characterized using SDQ-25 with the cutoff > 17
* Regular school attendence

Exclusion Criteria:

* IQ <80, ongoing psychiatric or psychotherapeutic treatment with regular appointments (at least once a month).

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Student's well-being and level of participation | T2 (baseline) vs. T3 (post intervention assessment within one week); T2 (baseline) vs. T4 (3 months follow-up)
  Student's well-being and level of participation measured by KIDSCREEN-27.

SECONDARY OUTCOMES:
Reduction of psychiatric burden | T2 (baseline) vs. T3 (post intervention assessment within one week); T2 (baseline) vs. T4 (3 months follow-up)
  Reduction of psychiatric burden as measured by SDQ-25, children/parent/teacher ) as well as SYMPTOM MONITORING as a daily individual symptom estimation on the likert scale in the Appversions.
Reduction of children's global impairment | T2 (baseline) vs. T3 (post intervention assessment within one week); T2 (baseline) vs. T4 (3 months follow-up)
  Reduction of children's global impairment will be assessed by the the German version of the Chil-dren Global Assessment Scale.
Feasibility measures | T2 (baseline) vs. T3 (post intervention assessment within one week); T2 (baseline) vs. T4 (3 months follow-up)
  Feasibility measures: number of students completed the programme, number of counselling ses-sions a student/parent, number of days/hours with STEPS support e.c..

OTHER OUTCOMES:
Determinants and mediators | T2 (baseline)
  Acceptance of the App (UTAUT Questionnaire & Questionnaire according to the Theory of Planned Behavior)
Determinants and mediators | T2 (baseline)
  Satisfaction with the program (ZUF-8 Zufriedenheitsfragebogen)
Determinants and mediators | T2 (baseline)
  Resilience of children (RS-13)
Determinants and mediators | T2 (baseline)
  Burden of parents (Parental Stress Scale)
Determinants and mediators | T2 (baseline)
  Burden of parents (ENRICHD-social support instrument)
Determinants and mediators | T2 (baseline)
  IQ (CFT 6-20R)
Health economic aspects | T4 (3 months follow-up)
  The assessment of psychosocial and health care service use (as a basis for the estimation of treatment costs for the parents) will be performed by the German version of the Client Socioeconomic and Services Receipt Inventory (CSSRI-DE)
Semi-structured interviews in the target populations | T4 (3 months follow-up)
  Semi-structured interviews in the target populations (patients, families, teachers, and health profes-sionals) will cover opinions, expectations, worries, beliefs, perceived benefits, risks, harms and dangers of the App, prevention programme, and digital literacy training. Particular attention will be paid to how target populations evaluate the introduction of the blinded-care treatment, and what benefits and problems they observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Child and Adolescent Psychiatry, RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dallinger VC, Krishnamoorthy G, du Plessis C, Pillai-Sasidharan A, Ayres A, Waters L, Groom Y, Alston O, Anderson L, Burton L. Utilisation of Digital Applications for Personal Recovery Amongst Youth with Mental Health Concerns. Int J Environ Res Public Health. 2022 Dec 14;19(24):16818. doi: 10.3390/ijerph192416818. PMID 36554700
- [Background] Damian AJ, Gallo JJ, Mendelson T. Barriers and facilitators for access to mental health services by traumatized youth. Child Youth Serv Rev. 2018 Jan;85:273-278. doi: 10.1016/j.childyouth.2018.01.003. Epub 2018 Jan 7. PMID 29795708
- [Background] Grist R, Porter J, Stallard P. Mental Health Mobile Apps for Preadolescents and Adolescents: A Systematic Review. J Med Internet Res. 2017 May 25;19(5):e176. doi: 10.2196/jmir.7332. PMID 28546138
- [Background] Heflinger CA, Hinshaw SP. Stigma in child and adolescent mental health services research: understanding professional and institutional stigmatization of youth with mental health problems and their families. Adm Policy Ment Health. 2010 Mar;37(1-2):61-70. doi: 10.1007/s10488-010-0294-z. PMID 20232133
- [Background] Iskra W, Deane FP, Wahlin T, Davis EL. Parental perceptions of barriers to mental health services for young people. Early Interv Psychiatry. 2018 Apr;12(2):125-134. doi: 10.1111/eip.12281. Epub 2015 Oct 20. PMID 26487568
- [Background] Punukollu M, Marques M. Use of mobile apps and technologies in child and adolescent mental health: a systematic review. Evid Based Ment Health. 2019 Nov;22(4):161-166. doi: 10.1136/ebmental-2019-300093. Epub 2019 Jul 29. PMID 31358537